CLINICAL TRIAL: NCT02662166
Title: Magnetic Resonance Imaging of Bladder Cancer
Brief Title: MRI in Clinical Staging and Estimation of Treatment Response in Bladder Cancer
Acronym: MIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Peter Boström, MD, PhD, Deah of Department, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6/1801/2014
Record Dates: First submitted 2015-01-05; First posted 2016-01-25 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; MRI; TUR-BT; cystectomy; chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI and biomarkers in bladder cancer (Experimental): Utilization of MR-imaging and biomarkers to stage bladder cancer and in estimation of chemosensitivity
  Interventions: Device: MR imaging

INTERVENTIONS:
Device: MR imaging — 3 T MRI of the urinary bladder

SUMMARY:
Bladder cancer (BC) as the most common malignancy arising from the urinary tract continues to be a major health problem. This prospective non-randomized study will enroll 150 patients undergoing magnetic resonance imaging (MRI) at different stages of their diagnostic and therapeutical process. The enrolled patients with suspected BC (BC) based on cystoscopy will have their initial MRI examination before transurethral resection of bladder tumor (TUR-BT) and biomarker collection. After pathology review of the histological specimens, patients will be treated according to standard clinical practice. The second MRI examination will be performed before therapeutic intervention, if TUR-BT alone is not sufficient enough. Neoadjuvant chemotherapy will be applied in high risk patients having muscle invasison, while intermediate risk patient - T1 high grade or carcinoma in situ patients - will be treated using Bacillus Calmette-Guerin (BCG) instilliations. After the completion of the neoadjuvant chemotherapy or BCG treatment, the patients will undergo the third MRI examination. Low risk patients will be followed by annual with MRI examination.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 85 years old
* Suspected BC based on cystoscopical evaluation.
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethical Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* History of serious cardiovascular, liver or kidney disease
* Uncontrolled serious infection
* Contraindications for MRI (cardiac pacemaker, intracranial clips etc)
* Patient refusing radical cystectomy or chemotherapy or BCG
* Intravesical Bacillus Calmette-Guerin instillations within 6 months before the first MRI examination

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of the multiparametric MRI (anatomical MRI, DCE-MRI, DWI) in the staging of bladder cancer | 24 months
  The accuracy of multiparametric MRI (anatomical MRI, DCE-MRI, DWI) in the staging of bladder cancer will be evaluated using transurethral resection of bladder tumor and cystectomy specimens

SECONDARY OUTCOMES:
Prediction of response to neo-adjuvant chemotherapy and/or BCG treatment evaluated by multiparametric MRI (anatomical MRI, DCE-MRI, DWI) | 24 months
  The aim is to evaluate predictive power of multiparametric MRI for estimation neo-adjuvant chemotherapy and/or BCG treatment response. Multiparametric MRI will be performed before neo-adjuvant chemotherapy and/or BCG treatment and patients will be followed using standard clinical follow up and/or undergo cystectomy.

OTHER OUTCOMES:
Estimation of chemosensitivity | 24 months
  Prevalence of patients responding neo-adjuvant chemotherapy, compared with the non-responders as evaluated by cystectomy specimens, according to various biomarkers and ex vivo tissue culturing will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Boström, MD, PhD, Principal Investigator — Department of Urology, University of Turku and Turku University Hospital
Locations (2):
- Finland (2):
  - Department of Urology, Central Hospital of Pori, Pori
  - University of Turku, Turku

REFERENCES:
- [Derived] Nikulainen I, Salminen AP, Jambor I, Merisaari H, Tammilehto V, Taimen P, Seikkula H, Bostrom PJ. Visual MRI T-category versus VI-RADS evaluation from multiparametric MRI in the detection of muscle-invasion in patients with suspected bladder cancer: single centre registered clinical trial (MIB-trial). Scand J Urol. 2021 Oct;55(5):354-360. doi: 10.1080/21681805.2021.1971290. Epub 2021 Aug 27. PMID 34448679